CLINICAL TRIAL: NCT03542305
Title: A PHASE 1, SINGLE DOSE OPEN-LABEL STUDY TO EVALUATE THE PHARMACOKINETICS OF LORLATINIB IN SUBJECTS WITH IMPAIRED RENAL FUNCTION
Brief Title: Lorlatinib Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: B7461010; RENAL IMPAIRMENT (Other: Alias Study Number)
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild (Experimental): Mild renal impairment
  Interventions: Drug: Lorlatinib
- Moderate (Experimental): Moderate renal impairment
  Interventions: Drug: Lorlatinib
- Severe (Experimental): Severe renal impairment
  Interventions: Drug: Lorlatinib
- Normal (Other): Normal renal function
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib single oral dose

SUMMARY:
This is a Phase 1, open-label, multi-center, single treatment study in subjects with normal renal function and varying degrees of renal impairment.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multi-center, single treatment study in subjects with normal renal function and varying degrees of renal impairment. Each subject will receive a single oral dose of lorlatinib administered in the fasted state. Subjects with mild, moderate, and severe renal impairment will be enrolled and normal healthy subjects will be enrolled as matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of non-childbearing potential
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Demonstrate stable renal function

Exclusion Criteria:

* Renal allograft recipients
* Any condition possibly affecting drug absorption (eg, gastrectomy)
* A positive urine drug test
* History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Screening supine triplicate 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec
* Second-degree or third-degree AV block (unless paced) or baseline PR interval >180 msec at any time prior to dosing of study treatment.
* Abnormalities in clinical laboratory tests at screening
* Pregnant or breastfeeding female subjects
* History of HIV, Hepatitis B, Hepatitis C, HIT, sensitivity to heparin
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Prism Clinical Research, LLC, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lin S, Gong J, Canas GC, Winkle P, Pelletier K, LaBadie RR, Ginman K, Pithavala YK. A Phase I Study to Evaluate the Pharmacokinetics and Safety of Lorlatinib in Adults with Mild, Moderate, and Severe Renal Impairment. Eur J Drug Metab Pharmacokinet. 2022 Mar;47(2):235-245. doi: 10.1007/s13318-021-00747-4. Epub 2022 Jan 11. PMID 35018553
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The mild renal impairment participants were recruited first. After lorlatinib was tolerated in at least 3 mild impairment participants, moderate impairment participants were enrolled. After dosing of 3 moderate impairment participants for at least 1 week, the remaining moderate impairment participants and the severe impairment participants were enrolled. The enrollment of normal renal function participants began after all renal impairment participants completed the PK collection.
Groups:
- Normal Function: Participants with normal renal function received a 100 mg single oral dose of lorlatinib tablet on day 1 with approximately 240 mL of ambient temperature water at approximately 0800 hours (±3 hours) following an overnight fast of at least 10 hours.
- Mild Impairment: Participants with mild renal impairment received a 100 mg single oral dose of lorlatinib tablet on day 1 with approximately 240 mL of ambient temperature water at approximately 0800 hours (±3 hours) following an overnight fast of at least 10 hours.
- Moderate Impairment: Participants with moderate renal function received a 100 mg single oral dose of lorlatinib tablet on day 1 with approximately 240 mL of ambient temperature water at approximately 0800 hours (±3 hours) following an overnight fast of at least 10 hours.
- Severe Impairment: Participants with severe renal function received a 100 mg single oral dose of lorlatinib tablet on day 1 with approximately 240 mL of ambient temperature water at approximately 0800 hours (±3 hours) following an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Started | 8 | 8 | 8 | 5
Completed | 8 | 8 | 8 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were randomized.
Groups:
- Normal Function: Participants with normal renal function received a 100 mg dose of lorlatinib tablets with approximately 240 mL of ambient temperature water at approximately 0800 hours (±3 hours) following an overnight fast of at least 10 hours.
- Total: Total of all reporting groups
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 5 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (3.66) | 59.0 (7.27) | 63.1 (4.88) | 60.4 (11.08) | 59.7 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 1 | 12
  Male | 5 | 5 | 3 | 4 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 5 | 7 | 8 | 3 | 23
  Black or African American | 3 | 0 | 0 | 2 | 5
  Asian | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Lorlatinib
Description: AUCinf was calculated by AUClast + (Clast*/kel), where AUClast was the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration; Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
ng*hr/mL | 8329 (33) | 8683 (29) | 9890 (27) | 11760 (37)
Statistical Analysis 1: Comparison: Normal Function vs Mild Impairment; Test type: Other; ANOVA; The natural log transformed parameter was used; Ratio (%) of Adjusted Geometric Means = 104.25, 90% CI 2-sided [79.73 to 136.31] — Normal renal function was the reference group. Mild renal impairment was test group. The estimate was derived from ratio (%) of adjusted geometric means of Test and Reference
Statistical Analysis 2: Comparison: Normal Function vs Moderate Impairment; Test type: Other; ANOVA; The natural log transformed parameter was used; Ratio (%) of Adjusted Geometric Means = 118.75, 90% CI 2-sided [91.43 to 154.24] — Normal renal function was the reference group. Moderate renal impairment was test group. The estimate was derived from ratio (%) of adjusted geometric means of Test and Reference
Statistical Analysis 3: Comparison: Normal Function vs Severe Impairment; Test type: Other; ANOVA; The natural log transformed parameter was used; Ratio (%) of Adjusted Geometric Means = 141.14, 90% CI 2-sided [97.82 to 203.66] — Normal renal function was the reference group. Severe renal impairment was test group. The estimate was derived from ratio (%) of adjusted geometric means of Test and Reference

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lorlatinib
Description: Cmax was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
ng/mL | 546.8 (48) | 549.7 (52) | 485.9 (24) | 504.8 (50)
Statistical Analysis 1: Comparison: Normal Function vs Mild Impairment; Test type: Other; ANOVA; The natural log transformed parameter was used; Ratio (%) of Adjusted Geometric Means = 100.53, 90% CI 2-sided [66.48 to 152.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Normal Function vs Moderate Impairment; Test type: Other; ANOVA; The natural log transformed parameter was used; Slope = 88.87, 90% CI 2-sided [64.18 to 123.06] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Normal Function vs Severe Impairment; Test type: Other; ANOVA; The natural log transformed parameter was used; Ratio (%) of Adjusted Geometric Means = 92.32, 90% CI 2-sided [56.58 to 150.63] — [estimate comment as in outcome 1, analysis 3]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a product or medical device; the event did not need to have a causal relationship with the treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and AEs. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Number of participants with both all-causality and treatment-related TEAEs are presented below.
Time Frame: Baseline up to 28 days after last dose of study treatment (approximately 29 days)
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
Participants
  All-causality AEs | 5 | 2 | 4 | 1
  All-causality SAEs | 0 | 0 | 0 | 0
  Treatment-related AEs | 3 | 2 | 1 | 1
  Treatment-related SAEs | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormalities
Description: The hematology, chemistry and urinalysis tests were included in the laboratory examination. Hematology evaluation included hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes, erythrocyte mean corpuscular volume, erythrocyte mean corpuscular hemoglobin concentration and erythrocyte mean corpuscular hemoglobin. Chemistry evaluation included blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid albumin, total protein, lipase and amylase. Urinalysis evaluation included decimal logarithm of reciprocal of hydrogen ion activity [pH], glucose, protein, blood, ketones, microscopy, ketones, nitrite, leukocyte esterase, urobilinogen, urine bilirubin and bacteria. The lab abnormalities were reported in accordance with the sponsor reporting standards.
Time Frame: Screening, Day -1, Day 2 and Day 6
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
Participants | 4 | 2 | 8 | 5

5. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Summarization Criteria
Description: Vital signs evaluations included supine diastolic blood pressure (DBP), and supine systolic blood pressure (SBP) were measured with the participant's arm supported at the level of the heart and recorded to the nearest mmHg after approximately 5 minutes of rest. Number of participants with vital signs data meeting the categorical summarization criteria is presented. The pre-specified criteria of vital signs data were categorized as follows: SBP (minimum) <90 mmHg, maximum of decrease and increase from baseline for SBP >=30 mmHg; DBP (minimum) <50 mmHg, maximum of decrease and increase from baseline for DBP>=20 mmHg.
Time Frame: Baseline up to 28 days after last dose of study treatment (approximately 29 days)
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
Participants
  Supine SBP < 90 mmHg | 0 | 1 | 0 | 0
  Supine SBP ≥ 30 mmHg increase | 0 | 0 | 2 | 1
  Supine SBP ≥ 30 mmHg decrease | 1 | 1 | 0 | 0
  Supine DBP < 50 mmHg | 0 | 1 | 0 | 0
  Supine DBP ≥ 20 mmHg increase | 0 | 0 | 1 | 1
  Supine DBP ≥ 20 mmHg decrease | 0 | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Categorical Summarization Criteria
Description: ECG evaluation included: PR interval, time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS interval), time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (QT interval), and QT interval corrected for heart rate using Fridericia's formula (QTcF interval). The pre-specified criteria of ESG data were categorized as below.
Time Frame: Screening, Day -1, 0 hours (pre-dose), 1 hour, 2 hours, 4 hours, 24 hours and 120 hours postdose.
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
Participants
  PR interval ≥ 200 to <220 msec | 0 | 0 | 0 | 1
  PR interval ≥ 200 to <240 msec | 0 | 0 | 0 | 0
  PR interval ≥ 240 to <260 msec | 0 | 0 | 0 | 0
  PR interval ≥ 260msec | 0 | 0 | 0 | 0
  QRS interval >120 msec | 0 | 0 | 0 | 0
  QT interval ≥ 500 msec | 0 | 0 | 0 | 0
  QTcF interval ≥ 450 to <480 msec | 0 | 0 | 0 | 0
  QTcF interval ≥ 480 msec | 0 | 0 | 0 | 0
  PR interval change from baseline ≥ 40 to <60 msec | 0 | 0 | 1 | 0
  PR interval change from baseline ≥ 60 to <80 msec | 0 | 0 | 0 | 0
  PR interval change from baseline ≥ 80 msec | 0 | 0 | 0 | 0
  PR interval percent change from baseline > 25% | 0 | 0 | 1 | 0
  QRS interval percent change from baseline ≥ 50% | 0 | 0 | 0 | 0
  QTcF interval change from baseline ≥ 30 to <60 msec | 0 | 0 | 0 | 0
  QTcF interval change from baseline ≥ 60 msec | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Lorlatinib
Description: AUClast was calculated by linear/Log trapezoidal method.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
ng*hr/mL | 8015 (32) | 8307 (28) | 8867 (24) | 10310 (36)

8. Other Pre Specified Outcome: Time for Cmax (Tmax) of Lorlatinib
Description: Tmax was observed directly from data as time of first occurrence.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
hours | 1.50 [1.00 to 4.00] | 1.00 [1.00 to 1.50] | 1.25 [1.00 to 4.00] | 1.00 [1.00 to 1.50]

9. Other Pre Specified Outcome: Terminal Elimination Plasma Half-life (t½) of Lorlatinib
Description: t1/2 was calculated by ln(2)/kel.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
hours | 25.64 (4.7500) | 28.08 (3.5156) | 39.40 (7.1019) | 41.66 (7.6081)

10. Other Pre Specified Outcome: Apparent Clearance After Oral Dose (CL/F) of Lorlatinib
Description: CL/F was calculated by Dose/AUCinf.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
L/hr | 12.02 (33) | 11.51 (29) | 10.11 (27) | 8.51 (37)

11. Other Pre Specified Outcome: Apparent Volume of Distribution Following Oral Dose (Vz/F) of Lorlatinib
Description: Vz/F was calculated by Dose/(AUCinf*kel). kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
L | 436.9 (24) | 462.9 (27) | 566.2 (21) | 503.8 (36)

12. Other Pre Specified Outcome: Renal Clearance (CLR) of Lorlatinib
Description: CLR was calculated by Ae/AUClast. Ae was cumulative amount of drug recovered unchanged in urine, which was calculated by sum of (urine concentration × sample volume) for each collection interval from 0 to time 120 hours postdose. Sample volume = (urine weight in g/1.020), where 1.020 g/mL is the approximate specific gravity of urine.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours postdose
Population: The analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 5
L/hr | 0.1095 (42) | 0.1382 (50) | 0.08199 (55) | 0.06872 (45)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study treatment (approximately 29 days)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Normal Function | Mild Impairment | Moderate Impairment | Severe Impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 5/8 | 2/8 | 4/8 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Function (N=8) | Mild Impairment (N=8) | Moderate Impairment (N=8) | Severe Impairment (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT03542305/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03542305/SAP_001.pdf